CLINICAL TRIAL: NCT06906861
Title: Epistaxis in Patients Receiving Oral Anticoagulants and Antiplatelet: Prevalence Risk Factors at a Tertiary Care Hospital in Nepal
Acronym: Epistaxis
Status: Completed | Type: Observational
Sponsor: Institute of medicine, Maharagjung medical campus (Other)
Responsible Party: Principal Investigator, Shiv Kumar Sah, Mr., Institute of medicine, Maharagjung medical campus
Other Study IDs: 263(6-11) E2, 080/081; 263(6-11) E2, 080/081 (Other: IOM)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Epistaxis
Keywords: Epistaxis, oral anticoagulants, antiplatelet, prevalence, risk factors, warfarin
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to determine the prevalence of epistaxis and identify the associated risk factors among patients receiving oral anticoagulants and antiplatelet at a tertiary care hospital in Nepal.

A cross-sectional study was conducted among 284 patients receiving oral anticoagulants at a tertiary care hospital over a one-year period. Data were collected through structured interviews and medical record reviews. The prevalence of epistaxis with corresponding 95% CI was calculated, and risk factors were analyzed using multivariate logistic regression. A receiver operating characteristic (ROC) curve was determined to establish the suitability of the model.

DETAILED DESCRIPTION:
Study Design and duration This study employed a hospital-based observational, cross-sectional design to determine the prevalence of epistaxis and identify the associated factors among patients on oral anticoagulants and antiplatelet medications at a tertiary care hospital in Nepal. The study was conducted at the department of emergency and ENT over a one-year period, from November 2023 to October 2024.

Study Setting and justification The study was conducted at the department of emergency and Ear Nose Throat (ENT) of Tribhuvan university teaching hospital (TUTH), Institute of Medicine (IOM), a tertiary care hospital of Nepal's premier healthcare institutions, situated in the heart of the capital city, Kathmandu. TUTH stands as the top referral hospital in the country and a public hospital in Kathmandu with 850 beds, which is recognized hospitals of Nepal with a good flow of patients from all over Nepal, making it easier to recruit a sufficient number of representing cases for the study. This hospital serves a diverse patient population across the country from both urban and rural areas, making an ideal setting for the representative samples to study on the prevalence and risk factors associated with epistaxis in patients taking anticoagulants and antiplatelet medications.

Study Population and selection criteria Inclusion and exclusion criteria The study included individuals aged 40 years or older who had been prescribed oral anticoagulants or antiplatelet agents for at least 3 months. Patients were excluded if they had a known bleeding disorder unrelated to the use of anticoagulant or antiplatelet medication, a history of coagulopathy or other bleeding disorders (e.g., hemophilia), recent craniofacial or nasal trauma or surgery within the past 6 months, a known history of nasal polyps or other nasal lesions, or if they declined to provide consent.

Variables of interest In this study, age, gender, residency, social habits, underlying medical conditions, types of anticoagulant and antiplatelet medications, and the duration of medication use were identified as exposure variables; whereas, the prevalence, severity, and frequency of epistaxis were evaluated as outcome variables.

Sample Size Determination

The sample size was determined using a Cochrane formula for cross-sectional studies (18):

N = Z2×P(1-P)

d2 where, Z is the Z-value corresponding to a 95% confidence level (1.96) P is the estimated prevalence of epistaxis in patients on anticoagulants/antiplatelet, based on previous, and d is the margin of error, set at 5%.

Assuming an estimated prevalence of epistaxis of 21% (19) and a 10% non-response rate, the final sample size was calculated to be 284 patients.

Sampling Method Patients were recruited through consecutive sampling from outpatient departments (ENT and Emergency) and inpatient wards. Recruitment continued until the calculated sample size was achieved.

Data Collection tool and technique Data were collected using a structured, pre-tested questionnaire administered through face-to-face interviews by trained research assistants, researcher and clinician involved in the study.

Data collection procedure:

The study initially identified potential participants from patients currently prescribed anticoagulant and antiplatelet medications who were visiting the ENT and Emergency Departments at TUTH. Informed consent was obtained from each participant prior to data collection. Socio-demographics including age, gender, occupation, place of residence, and lifestyle factors such as smoking and alcohol use were gathered. Relevant medical history was obtained from patient medical records, and, when necessary, interviews were conducted with patients or their relatives to gather information on comorbidities, history of epistaxis, frequency and severity of epistaxis, other bleeding episodes, and underlying medical conditions; Medication details, including Information on the types of medications and the duration of anticoagulant or antiplatelet therapy, which were obtained from medical and prescription records; clinical examination: A focused nasal examination was performed by an ENT specialist to assess for predisposing factors such as nasal septal deviation, mucosal dryness, and the presence of nasal polyps or other abnormalities Statistical Analysis Descriptive statistics were used to summarize the demographic and clinical characteristics of the study population. Continuous variables were expressed as means ± standard deviations (SD), while categorical variables were presented as frequencies and percentages. Bivariate analyses were conducted to explore associations between epistaxis and categorical variables using Chi-square tests or Fisher's exact tests, as appropriate, and independent t-tests or Mann-Whitney U tests were used for continuous variables. Variables with a p-value <0.05 in bivariate analysis were included in the logistic regression model. Crude and Adjusted odds ratios (AOR) with 95% confidence intervals (CI) were reported to identify the independent factors associated with the epistaxis. A p-value <0.05 was considered statistically significant in all analyses. All statistical analyses were conducted using SPSS, version 23 Ethical Considerations The study was approved by Institutional Review Committee (IRC- IOM), Institution of Medicine, Tribhuvan University prior to the commencement of the study. (Reference no. 263(6-11) E2, 080/081). Written informed consent was obtained from all participants before data collection. Confidentiality and privacy were ensured by anonymizing patient data and securing the database. Only the research team had access to the data. Patients who experienced active epistaxis during the study were provided with appropriate medical care, as per hospital protocol.

ELIGIBILITY:
Inclusion Criteria:

* The study included individuals aged 40 years or older who had been prescribed oral anticoagulants or antiplatelet agents for at least 3 months.

Exclusion Criteria:

* Patients were excluded if they had a known bleeding disorder unrelated to the use of anticoagulant or antiplatelet medication, a history of coagulopathy or other bleeding disorders (e.g., hemophilia), recent craniofacial or nasal trauma or surgery within the past 6 months, a known history of nasal polyps or other nasal lesions, or if they declined to provide consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The individuals aged 40 years or older who had been prescribed oral anticoagulants or antiplatelet agents for at least 3 months, admitted at the depart of ENT or Emergency at TUTH were the study population of the study
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Epistaxis in Patients Receiving Oral Anticoagulants and Antiplatelet: Prevalence Risk Factors at a Tertiary Care Hospital in Nepal | The study was conducted at the department of emergency and ENT over a one-year period, from November 2023 to October 2024.
  This study aims to determine the prevalence of epistaxis and identify the associated risk factors among patients receiving oral anticoagulants and antiplatelet at a tertiary care hospital in Nepal.

CONTACTS AND LOCATIONS:
Locations (1):
- IOM, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided